CLINICAL TRIAL: NCT07394673
Title: Postoperative Analgesic Efficacy of Ultrasound-Guided Serratus Posterior Superior Intercostal Plane Block in Arthroscopic Shoulder Surgery
Brief Title: Ultrasound-Guided Serratus Posterior Superior Intercostal Plane Block for Analgesia in Arthroscopic Shoulder Surgery
Acronym: SPSIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Merih Yıldız Eglen, Principal Investigator, MD, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BursaCityHOS 4
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain, Acute; Shoulder Pain; Serratus Posterior Superior Intercostal Plane Block
Keywords: postoperative analgesia; shoulder arthroscopy; serratus posterior superior intercostal plane block
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Active Comparator: Group SPSIP: Participants in this arm will receive an ultrasound-guided serratus posterior superior intercostal plane block before the surgery. Patients will be taken to the operating room after sensory and motor block assessment.
  Control group: No block procedures will be performed on patients in this arm. Both groups will receive general anesthesia using the standard anesthesia method; induction with lidocaine, propofol, fentanyl, and rocuronium. Maintenance will be provided by inhalation anesthesia and remifentanil infusion. Before the end of surgery, all patients will receive paracetamol, Tramadol, and Tenoxicam intravenously as standard postoperative analgesia.
  After surgery, patients will be extubated and taken to the post-anesthesia care unit. Patient-controlled analgesia devices will be attached to all patients in the post-anesthesia care unit.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SPSIP (Active Comparator): Group SPSIP Participants in this arm will receive an ultrasound-guided serratus posterior plane block .
  Interventions: Procedure: Group SPSIP: Serratus Posterior Superior İntercostal Plane Block (SPSIP)
- Group Control (No Intervention): No block procedures will be performed on patients in this arm

INTERVENTIONS:
Procedure: Group SPSIP: Serratus Posterior Superior İntercostal Plane Block (SPSIP) — Serratus Posterior Superior İntercostal Plane (SPSIP) Block will be performed before the surgery in seated position, under standard sterilization conditions.A linear ultrasound probe will be placed in the sagittal plane along the medial border of the scapula, and the second and third ribs, relevant muscles, and the pleura will be identified.
  The needle will be advanced into the interfascial plane between the serratus posterior superior and intercostal muscles. After confirmation with salin injection , the block will be performed by injecting 30 mL of 0.25% bupivacaine, and the cranio-caudal spread will be visualized under ultrasound.
  Arms: Group SPSIP

SUMMARY:
This study aimed to evaluate the effectiveness of serratus posterior superior intercostal plane (SPSIP) block in managing postoperative pain in patients undergoing arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Most patients undergoing arthroscopic shoulder surgery report pain in the postoperative period. Pain management remains a significant concern in patient management, as it affects surgical costs, postoperative mobility, length of hospital stay, patient satisfaction, and surgical outcomes. Multimodal analgesia is recommended for the management of postoperative pain. Regional analgesia is an important component of multimodal analgesia.

The serratus posterior superior intercostal plane (SPSIP) block is a novel regional analgesia technique described in 2023. SPSIP has been reported to provide near-complete sensory blockade in the posterior neck, shoulder, and hemithorax regions.

The main objective of this study is to investigate the effectiveness of SPSIP block in patients undergoing arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Classified as American Society of Anesthesiologists (ASA) physical status I-II-III
* Scheduled for elective shoulder arthroscopy surgery
* Surgery performed under general anesthesia
* Provision of written informed consent

Exclusion Criteria:

* Use of anticoagulant or antiplatelet medications
* Presence of bleeding diathesis or coagulation disorders
* Known allergy or hypersensitivity to local anesthetics or opioid medications
* Infection or history of previous surgery at the planned block site
* Alcohol or drug dependence
* Cognitive impairment preventing reliable pain assessment using the NRS
* Pregnancy or lactation
* Diabetes mellitus
* Renal or hepatic impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative 48-Hour PCA Opioid Consumption | Postoperative 0-8, 8-16, 16-24, 24-48 intervals
  Total amount of opioid delivered by the patient-controlled analgesia (PCA) device during the first 48 hours after surgery, recorded in milligrams(mg)

SECONDARY OUTCOMES:
QoR-15 Recovery Score | Postoperative 24th and 48th hours
  The investigators will use the Turkish version of Quality of Recovery (QoR) / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  Able to breathe easily Been able to enjoy food Feeling rested Have had a good sleep Able to look after personal toilet and hygiene unaided Able to communicate with Getting support from hospital doctors and nurses Able to return to work or usual home activities Feeling comfortable and in control Having a feeling of general well-being
  PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) Moderate pain Severe pain Nausea or vomiting Feeling worried or anxious Feeling sad or depressed
Dynamic and static NRS scores | 0, 2, 4, 8, 16, 24, and 48 hours postoperatively
  Numeric Rating Scale (NRS) (0-10 0: No pain 10: most pain felt) pain scores at rest or movement at predefined postoperative hours
Total rescue analgesic dose | Postoperative 24th and 48th hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered as
Time of first request for rescue analgesia, | Postoperative 48-Hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered. The time will be recorded.
Length of Hospital Stay | the day of surgery, the day of discharge from the hospital
  Number of days spent in hospital after surgery
Block and Opioid-Related Adverse Effects and Complications | Postoperative 48-Hours
  Block- and opioid-related adverse effects and complications, including but not limited to local anesthetic toxicity, hematoma, infection, nerve injury, nausea, vomiting, pruritus, sedation, and respiratory depression, will be recorded
Perioperative Remifentanil infusion dose | Start time: Start of anesthesia administration End time: Termination of anesthesia administration
  The amount of remifentanil administered in micrograms during general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Merih Yıldız Eglen, MD, Principal Investigator — Bursa City Hospital
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avci O, Gundogdu O, Balci F, Tekcan MN, Ozbey M. Efficacy of serratus posterior superior intercostal plane block (SPSIPB) on post-operative pain and total analgesic consumption in patients undergoing video-assisted thoracoscopic surgery (VATS): A double-blinded randomised controlled trial. Indian J Anaesth. 2023 Dec;67(12):1116-1122. doi: 10.4103/ija.ija_589_23. Epub 2023 Dec 13. PMID 38343684
- [Background] Kulturoglu G, Altinsoy S, Ozguner Y, Cataroglu CK. Novel Serratus Posterior Superior Intercostal Plane Block Provided Satisfactory Analgesia after Breast Cancer Surgery: Two Case Reports. Turk J Anaesthesiol Reanim. 2024 Feb 28;52(1):33-35. doi: 10.4274/TJAR.2024.231431. PMID 38414179
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093